CLINICAL TRIAL: NCT06565949
Title: The Effect of Carer Training on Pressure Ulcers in Palliative Care Patients
Brief Title: The Effect of Carer Training on Pressure Ulcers in Palliative Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, FATOŞ UNCU, assistant professor, Firat University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FU-SBF-FU-04
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Public Health Nursing
Keywords: Palliative Care; Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomised experimental study with pretest-posttest control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education group (Experimental): Caregivers in the experimental group will be given a detailed and planned training programme on pressure sores.
  Interventions: Other: Education group; Other: control group
- Control group (No Intervention)

INTERVENTIONS:
Other: Education group — aregivers in the experimental group will be given a detailed and planned training programme on pressure sores. The trainings will be held in a total of four sessions, with twenty minutes in each session, two weeks apart.
  Other Names: C
  Arms: Education group
Other: control group — In the first stage of the study, the participants in the experimental and control groups were asked to complete the 'Introductory Information Form' and '' Pressure sore knowledge test' will be completed. In the second stage of the research, no intervention will be made to the caregivers in the control group, and in the last stage of the research, 'Pressure sore knowledge test' will be filled in as post-test data for all participants.
  Arms: Education group

SUMMARY:
The aim of this article is to examine the effect of the training of carers caring for palliative care patients on the prevention and management of pressure ulcers. In this context, how the training affects the level of knowledge and practices of the carers will be evaluated. The findings obtained will contribute to improving the quality of patient care by providing strategic recommendations for the improvement of palliative care services.

DETAILED DESCRIPTION:
Palliative care is an approach that improves the quality of life of patients and their families facing problems related to life-threatening diseases. This care model focuses on meeting the physical, psychological, social and spiritual needs of patients. . Pressure ulcers are one of the most common and serious problems in palliative care. Pressure ulcers are injuries occurring on the skin or soft tissue. They develop due to pressure on certain parts of the body over a long period of time. If not treated immediately, they may cause fatal complications. Pressure ulcers affect more than 1 in 10 adult patients admitted to hospital and are highly preventable.

Most palliative care patients cannot provide self-care. Therefore, caregivers are one of the most important determinants of the patient's health status. At this point, the knowledge and skill levels of carers who provide direct care to patients are of great importance. Increasing the level of knowledge and awareness of caregivers to prevent pressure ulcers is a critical strategy to prevent the formation of these wounds and to accelerate the healing of existing wounds. In a systematic review of thirty-one articles, it was stated that pressure ulcers significantly limit many aspects of an individual's well-being, including mental and physical health and quality of life. Therefore, caregivers should have adequate knowledge about practices to prevent bedsores.

The aim of this article is to examine the effect of the training of carers caring for palliative care patients on the prevention and management of pressure ulcers. In this context, how the training affects the level of knowledge and practices of the carers will be evaluated. The findings obtained will contribute to improving the quality of patient care by providing strategic recommendations for the improvement of palliative care services.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Being the sole informal caregiver of the palliative care patient
* Being able to use physical abilities such as sight and hearing
* No cognitive and communication problems

Exclusion Criteria:

* Palliative care patient is not the only informal caregiver
* Cognitive and communication problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Pressure Wound Knowledge Test | 2 month
  CBRT is a 3-point Likert type (true, false, don't know) questionnaire consisting of 17 questions prepared by the researchers in line with the literature. Five of the questions in the test were designed to be reverse scored and 12 were designed to be scored normally. The minimum score of the knowledge test is 0 and the maximum score is 17. The KR-20 value of this measurement tool was calculated as 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Fatoş Uncu, PhD, Principal Investigator — funcu@firat.edu.tr
Locations (1):
- Firat University, Elâzığ, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No